CLINICAL TRIAL: NCT01976793
Title: Retrospective Observational Study to Estimate the Duration of Initial Antidepressant Treatment in Patients With Recurrent Depressive Disorder Who Demonstrated a Suboptimal Response to Therapy: DIANA Study
Brief Title: Retrospective Observational Study DIANA Study
Acronym: DIANA
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-NRU-ATC-2013/1
Record Dates: First submitted 2013-10-24; First posted 2013-11-06 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Major Depressive Episode
Keywords: Recurrent depressive disorder; Depression; Depressive episode; Atypical antipsychotics
MeSH Terms: conditions — Depressive Disorder; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients with major depression: Inpatients and outpatients diagnosed with an episode of major depression relating to RDD (ICD-10, Version 2010) during the period from January 1, 2012 till September 30, 2013. Initially treated with antidepressant monotherapy, using a flexible dosage regimen if required, for at least 2 week

SUMMARY:
This Non-Interventional Study (NIS) is intended to evaluate the duration of treatment with an initial antidepressant taken as monotherapy in patients in whom treatment was changed because of suboptimal response at physician's discretion. This will address unmet medical needs of patients with a depressive episode related to RDD (ICD-10, Version 2010), who have failed to respond adequately to initial treatment with an antidepressant and contribute to an understanding of the usual approaches that physicians adopt to monitor initial treatment efficacy in RDD (Recurrent Depressive Disorder). The study will also focus on second-line therapy in hard to treat patients, describing the different pharmacotherapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male aged between 18 and 65 years Inpatients and outpatients diagnosed with an episode of major depression relating to RDD (ICD-10, Version 2010) during the period from January 1, 2012 till September 30, 2013 3. Initially treated with antidepressant monotherapy, using a flexible dosage regimen if required, for at least 2 weeks 4. Initial treatment changed because of a suboptimal response at physician's discretion, which is clearly documented in the patient's medical chart.

Exclusion Criteria:

Patients currently participating in any other clinical or non-interventional trial, or have completed their participation with the last 30 days.

2. Patients with current psychiatric or general medical conditions which require concomitant use of lithium, thyroid hormones, or atypical antipsychotics 3. Patients with unstable general medical condition. 4. Patients who were pregnant or were suspected to be pregnant during the period when a patient had received treatment for MDE (Major Depressive Episode).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Inpatients and outpatients diagnosed with an episode of major depression relating to RDD (ICD-10, Version 2010) during the period from January 1, 2012 till September 30, 2013. Initially treated with antidepressant monotherapy, using a flexible dosage regimen if required, for at least 2 weeks
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2013-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Duration of treatment considered as time between initiation of antidepressant monotherapy and the alteration and/or augmentation of pharmacotherapy | up to 6 months
  Primary objective: The primary objective of this NIS is to evaluate the duration of treatment with an initial antidepressant taken as monotherapy in patients in whom treatment was changed because of suboptimal response at physician's discretion.

SECONDARY OUTCOMES:
Pharmacotherapy strategy for the second line treatment | up to 6 months
  Distribution of the various pharmacotherapy strategies following suboptimal response: (switch; augmentation; combination of switch and augmentation and discontinuation of pharmacotherapy) among the patients population.
International Non-Proprietary Name (INN) of pharmacological agents prescribed for augmentation | Up to 6 months
  Rate of the different pharmacological agents prescribed for augmentation; rout of their administration; mean and median duration of courses of treatment
Doses of pharmacological agents used for augmentation | Up to 6 months
  Mean and median doses of pharmacological agents used for augmentation
Source of the patient's referral to a psychiatrist | up to 6 months
  Distribution of various sources of the patient's referral to a psychiatrist (psychotherapist; neurologist; internist; physician of other speciality; psychologist; came himself; other; and not known

CONTACTS AND LOCATIONS:
Overall Officials: Alla Avedisova, Prof, Principal Investigator — Center of Social and Forensic Psychiatry, Moscow; Karin Otter, PhD, Study Director — AstraZeneca Russia; Anatoly Smulevich, Prof, Principal Investigator — Scientific centef of Mental Health, Moscow; Galina Mazo, Prof, Principal Investigator — St Petersburg Scientific Psyconeurology institute
Locations (8):
- Russia (8):
  - Research Site, Ivanovo
  - Research Site, Kazan'
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Rostov-on-Don
  - Research Site, Saint Petersburg
  - Research Site, Stavropol
  - Research Site, Yaroslavl

REFERENCES:
- See also: NIS-NRU-ATC-2013/1 Clinical Study Report Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1913&filename=NIS-NRU-ATC-2013-1_Clinical_Study_Report_Synopsis.pdf